CLINICAL TRIAL: NCT00534105
Title: Study of Lipid Metabolism in Gestational Diabetes
Brief Title: Lipid Metabolism in Gestational Diabetes
Status: Completed | Type: Observational
Sponsor: Baystate Medical Center (Other)
Responsible Party: Principal Investigator, Glenn Markenson, Director, Maternal Fetal Medicine, Baystate Medical Center
Other Study IDs: IRB07-121
Record Dates: First submitted 2007-09-21; First posted 2007-09-24 (Estimated); Results first posted 2013-09-11 (Estimated); Last update posted 2013-09-11 (Estimated); Status verified 2013-07

CONDITIONS: Gestational Diabetes; Hyperlipidemia
Keywords: Pregnancy; Gestational diabetes; Hyperlipidemia
MeSH Terms: conditions — Diabetes, Gestational; Hyperlipidemias | interventions — Cholesterol; Triglycerides

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Gestational Diabetics: Patients with Gestational Diabetes
  Interventions: Other: Total Cholesterol; Other: Triglyceride; Other: HDL; Other: LDL
- 2: Normal pregnant women without gestational diabetes
  Interventions: Other: Total Cholesterol; Other: Triglyceride; Other: HDL; Other: LDL

INTERVENTIONS:
Other: Total Cholesterol
Other: Triglyceride
Other: HDL
Other: LDL

SUMMARY:
The purpose of this pilot study is to determine if, during pregnancy, women with GDM have an exaggerated lipid response compared to non-gestational diabetics. If a difference is noted, further studies will explore the possibility of screening gestational diabetics during their pregnancy for hyperlipidemia to determine if prenatal screening can predict postpartum risk for hyperlipidemia. In addition the relationship, if any between maternal lipid dysfunction and placental disease will be explored.

This will be a prospective cohort study. As part of routine prenatal care, women receive a one hour glucose challenge test to screen for gestational diabetes. Those women with elevated values then require a three hour glucose tolerance test, which is a diagnostic test for gestational diabetes. All women that are scheduled to receive a three hour GTT will be identified and ask to enroll in this study. 46 women whose three hour GTT is normal and thus do not have GDM, will be compared to 46 women with an abnormal three hour GTT and thus would have the diagnosis of GDM. Enrolled women will have a lipid panel consisting of; total cholesterol, triglycerides, HDL and LDL cholesterol at the time of their fasting glucose blood sample. In addition, a repeat lipid panel will be sent at the time of the third hour sample, to assess changes, if any due to the glucose challenge. Umbilical cord blood samples will be sent in order to obtain newborn lipid profiles. Women in both the GDM and normal groups will be asked to return 6-8 weeks

DETAILED DESCRIPTION:
The purpose of this pilot study is to determine if, during pregnancy, women with GDM have an exaggerated lipid response compared to non-gestational diabetics. If a difference is noted, further studies will explore the possibility of screening gestational diabetics during their pregnancy for hyperlipidemia to determine if prenatal screening can predict postpartum risk for hyperlipidemia. In addition the relationship, if any between maternal lipid dysfunction and placental disease will be explored. Subsequent studies could also explore the possible perinatal complications associated with elevated lipids and or metabolic syndrome.

C. Experimental Design, Methodology and Expected Results

Study Design:

We propose a prospective cohort design.

Study Population:

All women that are scheduled to receive a three hour GTT to rule out gestational diabetes would be identified and ask to enroll in this study. Specifically, eligible patients will be women who failed their glucose challenge test (GCT) and are scheduled for the follow-up three hour glucose tolerance test (GTT). The GCT is routinely performed among all prenatal care patients at 24-28 wks gestation. The 3 hour GTT requires patients to be fasting overnight. A fasting blood glucose is sampled, and the patients are given a 100 gram glucose drink. Serum glucose samples are then taken at one, two and three hours after the glucose loading. The "exposed" group will be defined as women diagnosed with GDM (elevated glucose values on two or more samples in the three hour GTT). The "unexposed" group will be defined as women with no abnormal glucose values in the three hour GTT.

ELIGIBILITY:
Inclusion Criteria:

* Pregnancy
* Abnormal one hour glucose challenge test
* "Normal" controls group one hour test between 135 mg% and 150 mg%
* "Gestational diabetic" group with two abnormal values on a 3 hour GTT

Exclusion Criteria:

* History of diagnosis of diabetes, hypertension, heart disease or chronic renal disease
* Prior history of lipid disorder or metabolic syndrome
* Current medications thought to adversely influence glucose tolerance (i.e. prednisone or other steroids and systemic beta-mimetic drugs)
* Non-singleton pregnancy
* < 16 years of age or over 40 years of age
* Not planning to deliver at Baystate Medical Center
* Twins

Ages: 16 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pregnant women
Sampling Method: Non-Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2007-09; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Glenn R Markenson, MD, Principal Investigator — Baystate Medical Center
Locations (1):
- Baystate Medical Center, Springfield, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Pregnant patients presenting for gestational diabetes screening
Pre-assignment Details: Only uncomplicated obstetrical patients
Groups:
- Gestational Diabetics: Patients with Gestational Diabetes with a lipid screening performed during the pregnancy.
- Normal Pregnancies: Normal pregnant women without gestational diabetes
Period: Overall Study
Arm/Group | Gestational Diabetics | Normal Pregnancies
Started | 47 | 59
Completed | 24 | 20
Not Completed | 23 | 39
Not completed — Lost to Follow-up | 23 | 39

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Gestational Diabetics | Normal Pregnancies | Total
Number analyzed (Participants) | 47 | 59 | 106
Age Continuous [Median (Inter-Quartile Range); unit: years]
  Age at Recruitment | 32 [30 to 36] | 30 [26 to 34] | 31 [28 to 35]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 59 | 106
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 47 | 59 | 106

OUTCOME MEASURES:

1. Primary Outcome: Cholesterol
Description: Cholesterol values were obtained at least 6 weeks postpartum from the gestational diabetic group and the normal controls
Time Frame: Postpartum
Measure: Mean (Inter-Quartile Range); unit: mg/dl
Arm/Group | Gestational Diabetics | Normal Pregnancies
Number analyzed (Participants) | 24 | 20
mg/dl | 204 [139 to 330] | 201 [169 to 228]

2. Secondary Outcome: Triglyceride Values
Description: Triglyceride values were obtained at least 6 weeks postpartum in both the gestational diabetic group and the normal controls.
Time Frame: Postpartum
Measure: Mean (Inter-Quartile Range); unit: mg/dl
Arm/Group | Gestational Diabetics | Normal Pregnancies
Number analyzed (Participants) | 24 | 20
mg/dl | 118 [74 to 174] | 83 [52 to 109]

3. Secondary Outcome: HDL
Description: as for outcome 2
Time Frame: Postpartum
Measure: Mean (Inter-Quartile Range); unit: mg/dl
Arm/Group | Gestational Diabetics | Normal Pregnancies
Number analyzed (Participants) | 24 | 20
mg/dl | 51 [41 to 57] | 57 [52 to 69]

4. Secondary Outcome: LDL
Description: LDL values were obtained at least 6 weeks postpartum in both the gestational diabetic group and the normal controls.
Time Frame: Postpartum
Measure: Mean (Inter-Quartile Range); unit: mg/dl
Arm/Group | Gestational Diabetics | Normal Pregnancies
Number analyzed (Participants) | 24 | 20
mg/dl | 124 [110 to 154] | 120 [83 to 150]

ADVERSE EVENTS:
Arm/Group | Gestational Diabetics | Normal Pregnancies
Serious Adverse Events (participants affected / at risk) | 0/47 | 0/59
Other Adverse Events (participants affected / at risk) | 0/47 | 0/59

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes